CLINICAL TRIAL: NCT02960867
Title: European Registry of Dialysis Treatment of Pediatric Acute Kidney Injury (AKI)
Acronym: EurAKID
Status: Completed | Type: Observational
Sponsor: Mariella Enoc (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor-Investigator, Mariella Enoc, Principal Investigator, Bambino Gesù Hospital and Research Institute
Organization: Bambino Gesù Hospital and Research Institute (Other)
Other Study IDs: 1041_OPBG_2016
Record Dates: First submitted 2016-11-04; First posted 2016-11-10 (Estimated); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Acute Kidney Injury
Keywords: paediatric; kidney
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute kidney injury (AKI) is a frequent clinical condition in hospitalized, in particular, in critically ill children. Moreover, AKI is an independent predictor of mortality. An incidence of AKI in pediatric intensive care units (PICU) between 10 and 62% has been reported in recent clinical trials adopting pRIFLE or AKIN criteria, with the highest risk present in cardiac surgery patients. Despite significant developments in the management of AKI, the overall mortality rate of patients with AKI has not improved significantly. Currently, there is no consensus concerning the optimum dialysis modalities to adopt in pediatric AKI. No studies have prospectively compared the efficacy of different types of RRT for pediatric AKI. While PD remains the most commonly used modality in children worldwide, over the last decade CRRT has become the preferred treatment modality for critically ill children with AKI in North America.

The investigators have recently conducted a survey among 34 European Pediatric Nephrology Centers in the ESCAPE Network to obtain current information on dialysis management practices in children. Approximately 900 children with AKI requiring dialysis are managed at these 34 centers per year. This number supports the creation of a prospective European AKI registry.

DETAILED DESCRIPTION:
The main scope of the Registry is to report the epidemiology and outcome of children with AKI treated with dialysis in over 30 Pediatric Nephrology Centers in Europe. Secondary aims are to verify the association of a specific dialysis modality with the outcome and the association of primary disease, co-morbidities, nephrotoxic agents, fluid overload, anuria, basic hemodynamic parameters (BP, HR), basic nutritional intakes (protein and calorie supply) with the outcome.

Data capture will be exclusively web-based via electronic case report forms. Every participating site will be provided with a unique code and password that identify the corresponding site.

ELIGIBILITY:
Inclusion Criteria:

* Children with AKI at Hospital admission or who developed AKI during hospitalization treated with dialysis (PD, HD, CRRT)
* Age: 0-18 yrs

Exclusion Criteria:

* Children with known preexisting CKD (i.e.: AKI on CKD)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with AKI admitted to general PICUs and to cardiac ICUs will be included in the Registry.
Sampling Method: Probability Sample
Enrollment: 1892 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
incidence of AKI requiring dialysis in PICU and non-PICU children | 3 years
  urine output and serum creatinine

SECONDARY OUTCOMES:
Mortality rates | 3 years
  mortality
difference in mortality related to dialysis modality | 3 years
  CRRT modality (CVVH, CVVHD, CVVHDF)
difference in the primary outcome related to duration of mechanical ventilation | 3 years
  duration of mechanical ventilation
difference in the primary outcome related to severity score | 3 years
  severity score
difference in the primary outcome related to SpO2 | 3 years
  SpO2
difference in the primary outcome related to FiO2 | 3 years
  FiO2
difference in the primary outcome related to Mean Airway Pressure | 3 years
  Mean Airway Pressure
difference in the primary outcome related to paO2 | 3 years
  paO2

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Picca, Study Chair — Bambino Gesù Children's Hospital; Isabella Guzzo, Principal Investigator — Bambino Gesù Children's Hospital
Locations (1):
- Department of Nephrology-Urology "Bambino Gesù" Children's Research Hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schneider J, Khemani R, Grushkin C, Bart R. Serum creatinine as stratified in the RIFLE score for acute kidney injury is associated with mortality and length of stay for children in the pediatric intensive care unit. Crit Care Med. 2010 Mar;38(3):933-9. doi: 10.1097/CCM.0b013e3181cd12e1. PMID 20124891
- [Result] Bailey D, Phan V, Litalien C, Ducruet T, Merouani A, Lacroix J, Gauvin F. Risk factors of acute renal failure in critically ill children: A prospective descriptive epidemiological study. Pediatr Crit Care Med. 2007 Jan;8(1):29-35. doi: 10.1097/01.pcc.0000256612.40265.67. PMID 17251879
- [Result] Medina Villanueva A, Lopez-Herce Cid J, Lopez Fernandez Y, Anton Gamero M, Concha Torre A, Rey Galan C, Santos Rodriguez F. [Acute renal failure in critically-ill children. A preliminary study]. An Pediatr (Barc). 2004 Dec;61(6):509-14. doi: 10.1016/s1695-4033(04)78437-4. Spanish. PMID 15574251
- [Result] Akcan-Arikan A, Zappitelli M, Loftis LL, Washburn KK, Jefferson LS, Goldstein SL. Modified RIFLE criteria in critically ill children with acute kidney injury. Kidney Int. 2007 May;71(10):1028-35. doi: 10.1038/sj.ki.5002231. Epub 2007 Mar 28. PMID 17396113
- [Result] Basu RK, Zappitelli M, Brunner L, Wang Y, Wong HR, Chawla LS, Wheeler DS, Goldstein SL. Derivation and validation of the renal angina index to improve the prediction of acute kidney injury in critically ill children. Kidney Int. 2014 Mar;85(3):659-67. doi: 10.1038/ki.2013.349. Epub 2013 Sep 18. PMID 24048379
- [Result] Barrantes F, Tian J, Vazquez R, Amoateng-Adjepong Y, Manthous CA. Acute kidney injury criteria predict outcomes of critically ill patients. Crit Care Med. 2008 May;36(5):1397-403. doi: 10.1097/CCM.0b013e318168fbe0. PMID 18434915
- [Result] Duzova A, Bakkaloglu A, Kalyoncu M, Poyrazoglu H, Delibas A, Ozkaya O, Peru H, Alpay H, Soylemezoglu O, Gur-Guven A, Bak M, Bircan Z, Cengiz N, Akil I, Ozcakar B, Uncu N, Karabay-Bayazit A, Sonmez F; Turkish Society for Pediatric Nephrology Acute Kidney Injury Study Group. Etiology and outcome of acute kidney injury in children. Pediatr Nephrol. 2010 Aug;25(8):1453-61. doi: 10.1007/s00467-010-1541-y. Epub 2010 May 30. PMID 20512652
- [Result] Alkandari O, Eddington KA, Hyder A, Gauvin F, Ducruet T, Gottesman R, Phan V, Zappitelli M. Acute kidney injury is an independent risk factor for pediatric intensive care unit mortality, longer length of stay and prolonged mechanical ventilation in critically ill children: a two-center retrospective cohort study. Crit Care. 2011 Jun 10;15(3):R146. doi: 10.1186/cc10269. PMID 21663616
- [Result] Alabbas A, Campbell A, Skippen P, Human D, Matsell D, Mammen C. Epidemiology of cardiac surgery-associated acute kidney injury in neonates: a retrospective study. Pediatr Nephrol. 2013 Jul;28(7):1127-34. doi: 10.1007/s00467-013-2454-3. Epub 2013 Mar 22. PMID 23519522
- [Derived] Guzzo I, de Galasso L, Bayazit AK, Yildizdas D, Schmitt CP, Hayes W, Shroff R, Jankauskiene A, Virsilas E, Longo G, Vidal E, Mir S, Bulut IK, Tkaczyk M, Mencarelli F, Bertulli C, Cvetkovic M, Kostic M, Paglialonga F, Montini G, Yilmaz E, Teixeira A, Atmis B, Schaefer F. Acute paediatric kidney replacement therapies in Europe: demographic results from the EurAKId Registry. Nephrol Dial Transplant. 2022 Mar 25;37(4):770-780. doi: 10.1093/ndt/gfab280. PMID 34586417